CLINICAL TRIAL: NCT07316647
Title: Using Conversational AI to Teach Growth Mindset Skills to Youths in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, John Weisz, Henry Ford II Research Professor of the Social Sciences, Department of Psychology, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0827
Record Dates: First submitted 2025-12-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Youth Mental Health; Anxiety; Depression
Keywords: growth mindset; brief digital mental health intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Half the students will be randomly assigned to receive the full intervention at baseline, while the other half (control group) will complete a usual school assignment; after 7 weeks, the control group will receive a shortened (15-minute) version of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth mindset training (Experimental): Receives growth mindset training via 45-minute interaction with conversational AI
  Interventions: Behavioral: Growth mindset training using conversational AI
- Usual classroom activities (No Intervention): Performs usual classroom activities during the intervention period; receives delayed and shortened intervention at the conclusion of the study

INTERVENTIONS:
Behavioral: Growth mindset training using conversational AI — Participants will interact with an AI chatbot for approximately 45 minutes. The tutorial has a structured script and pauses at section boundaries to allow for brief interactions. It also contains culturally-grounded comics and illustrations with role-playing scenarios to engage with students.
  Arms: Growth mindset training

SUMMARY:
This study aims to test whether a brief digital intervention using conversational AI can improve mental health outcomes among school-aged youth (grades 6-8) in India, where most young people with mental health issues do not receive treatment. The intervention teaches "growth mindset", the belief that skills and abilities can improve with effort, via a 45-minute interactive conversation with an AI chatbot (spread across two class periods). A randomized controlled trial with approximately 430 students at a private, English-medium school in Bangalore will evaluate whether interacting with the chatbot can reduce symptoms of anxiety and depression while enhancing growth mindset beliefs. Half the students will receive the full intervention at baseline, while the other half (control group) will complete a usual school assignment; after 7 weeks, the control group will receive a shortened (15-minute) version of the growth mindset intervention. Participants will complete 10-minute surveys at baseline, 3 weeks, and 7 weeks, after which all students will receive a printed booklet with all the information from the chatbot. This study represents one of the first randomized controlled trials evaluating conversational AI as a brief digital intervention for youth mental health.

DETAILED DESCRIPTION:
Globally, 300 million youths have a diagnosable mental disorder and more reside in India than any other country. Yet, in India, where this study is based, most youths affected by mental health issues do not receive treatment. Symptoms are especially prevalent during high school, when many students show signs of depression and anxiety. Given myriad challenges in accessing mental healthcare, some have turned to conversational AIs such as ChatGPT and Claude for personalized support. However, there are few rigorous tests of whether such tools can improve mental health.

This study aims to bridge this gap by combining conversational AI with evidence-based intervention for youth mental health-specifically, a growth mindset intervention, which promotes the belief that abilities are not innate but can be improved with effort. It is well known that growth mindset interventions can improve academic performance. In addition, researchers have shown that brief, computer-guided growth mindset training can reduce symptoms of anxiety and depression that sustain 3-9 months post-intervention, and not only in the United States. However, until now, these interventions have been delivered via static, standardized websites that few people use.

The intervention considered is a 45-minute interactive lesson on growth mindset, embedded within a conversational AI. Similar to prior interventions, the content includes modules on understanding growth mindset, its basis in neuroplasticity, and roleplaying scenarios. Each module includes interactive discussions with the AI (e.g., "in your words, what is a growth mindset?", "in the above scenario, how could a growth mindset apply?")

The specific aim of the study is to test whether a brief, AI-enabled growth mindset intervention offers measurable benefits for school-aged youth in India. A randomized controlled trial with about 430 students (grades 6-8) will measure whether the AI-enabled training leads to changes in growth mindset beliefs and skills as well as symptoms of anxiety and depression, relative to a control group that receives a shortened intervention after 7 weeks. Brief, 10-minute questionnaires will be administered to all participants at baseline, 3 weeks, and 7 weeks. At the conclusion of the trial, all students will receive a printed booklet with content from the full intervention. The study will take place in an English-medium private school in Bangalore, India, which serves a diversity of students.

The growth mindset intervention may also benefit academic performance, and the school partner, at its discretion, may be able to integrate it into part of their standard curriculum following the completion of the study. However, the specific research question is whether the chatbot interaction yields measurable improvements in youth mental health. Given the preponderance of AI chatbots aiming to address various aspects of mental health, such measurement is as important as it is rare. This study will contribute to the growing evidence base on how technology can inform and support youth mental health.

ELIGIBILITY:
Inclusion Criteria:

* Youth in grades 6-8 at our partner school
* Youth assents to participate and a parent/guardian provides passive consent (does not opt-out of participation)

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Behavior and Feelings Survey - Internalizing Subscale (full sample) | Baseline, 3 weeks, 7 weeks
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing Subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms (BFS; Weisz et al., 2020).
Student Perceived Program Acceptability and Helpfulness | Immediately post-intervention
  Assessed via the Program Feedback Scale (Schleider et al., 2019). This scale consists of 7 items rated on a 1 to 5 scale, with higher scores indicating greater acceptability and helpfulness.

SECONDARY OUTCOMES:
Change in Behavior and Feelings Survey - Internalizing Subscale (elevated subsample) | Baseline, 3 weeks, 7 weeks
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing Subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms (BFS; Weisz et al., 2020).
Change in Growth Mindset Beliefs (full sample and elevated subsample) | Baseline, 3 weeks, 7 weeks
  Assessed via the Growth Mindset Scale (Sigmundsson & Haga, 2024), adapted to a lower reading level. This scale consists of 8 items, rated on a scale from 1 (not like me at all) to 5 (very much like me).
Growth mindset reflections (intervention group) | 3 weeks, 7 weeks
  Assessed with brief questions to check recall and use of growth mindset as well as intent to apply it in the future:
  * In one sentence, what is the main idea of growth mindset?
  * Have you used growth mindset for anything at school or home in the past few weeks? [Yes, Not yet, I'm not sure]
  * [If they answer "Yes"] Please share what happened. What did you do or think?
  * How might you use growth mindset in the next month? Be sure to explain: (i) WHAT you want to get better at. This could be a school subject, a skill, or any personal goal, (ii) HOW you will improve. This could include practicing, asking for help, or any of the tips above!

CONTACTS AND LOCATIONS:
Overall Officials: John R Weisz, Ph.D., Principal Investigator — Harvard University
Locations (1):
- Partner school, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
To respect concerns shared by our school partner regarding privacy of student data, individual participant data will not be shared with outside researchers.

REFERENCES:
- [Background] Weisz JR, Vaughn-Coaxum RA, Evans SC, Thomassin K, Hersh J, Ng MY, Lau N, Lee EH, Raftery-Helmer JN, Mair P. Efficient Monitoring of Treatment Response during Youth Psychotherapy: The Behavior and Feelings Survey. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):737-751. doi: 10.1080/15374416.2018.1547973. Epub 2019 Jan 18. PMID 30657721

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Version 1.0 (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT07316647/Prot_SAP_ICF_000.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Version 1.1 (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT07316647/Prot_SAP_ICF_001.pdf